CLINICAL TRIAL: NCT05675748
Title: A Non-interventional Real-world Study Evaluating the Efficacy and Safety of Azvudine in Nursing Home Patients With Mild/Normal COVID-19
Brief Title: Real-world Study Evaluating the Efficacy and Safety of Azvudine in Nursing Home Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Collaborators: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry); Huashan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FNC-Covid202
Record Dates: First submitted 2023-01-06; First posted 2023-01-09 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — azvudine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Azvudine — Azvudine tablets are taken orally 5mg daily for a maximum of 14 days

SUMMARY:
This study was a multicenter, non-intervention, real world study. To evaluate the efficacy and safety of azvudine in nursing homes with mild/common COVID-19 patients. The primary outcome measure was the proportion of patients with severe/critical illness within 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Living in a nursing home who has taken or intends to take azvudine tablets depending on their condition;
2. Mild/normal subjects who are SARS-CoV-2 RT-RCR positive or antigen-positive;
3. Subjects have at least one or more of the following clinical symptoms of COVID-19 in the 24 hours prior to initial administration, including but not limited to: fever, cough, sore throat, stuffy or runny nose, headache, muscle pain, nausea, vomiting, diarrhea, shortness of breath or difficulty breathing, chills or chills;
4. Volunteer to participate in the experiment and sign the informed consent in person or complete the informed consent over the phone.

Exclusion Criteria:

1. Subjects have received antiviral therapy, such as Paxlovid and SARS-CoV-2 monoclonal antibody therapy (except previous treatment for COVID-19 infection) before entering the study;
2. Shortness of breath, RR≥30 times/min or resting state, oxygen saturation of finger when sucking air ≤93%;
3. Mechanical ventilation is required or expected to be urgently required;
4. Severe infections requiring systemic treatment within 14 days prior to initial medication;
5. Use of other antiviral drugs (such as anti-HIV, hepatitis B, and hepatitis C drugs) within 14 days prior to the first medication.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: nursing homes patients with mild/common COVID-19 symptom
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with severe/critical illness within 28 days | up to 28 days from the first dose of Azvudine for treatment SARS-CoV-2 infection

SECONDARY OUTCOMES:
all-cause mortality within 28 days | up to 28 days from the first dose of Azvudine for treatment SARS-CoV-2 infection
Proportion of hospitalization within 28 days and the duration of hospitalization | up to 28 days from the first dose of Azvudine for treatment SARS-CoV-2 infection